CLINICAL TRIAL: NCT03646344
Title: Heme Arginate in Transplantation Study - a Multi-centre Blinded Parallel-group Randomised Trial of Heme Arginate Versus Placebo to Reduce Delayed Graft Function in Kidney Transplant Recipients
Brief Title: Heme Arginate in Transplantation Study
Acronym: HOT2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID
Sponsor: University of Edinburgh (Other)
Collaborators: Kidney Cancer UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC17065
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2021-06

CONDITIONS: Renal Transplant Rejection; Renal Transplant Failure
Keywords: Deceased donor renal transplantation; Heme Arginate; Delayed graft function
MeSH Terms: conditions — Delayed Graft Function | interventions — heme arginate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multi-centre, parallel group 1:1 randomised placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There will be an unblinded member of the research team (the individual administering the intervention) but otherwise the participant, the other members of the research team, the clinical team and blinded assessors will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Group (Active Comparator): Will receive Heme Arginate (IMP) at a dose of 3mg/kg over 30mins. Participants will receive infusions of the IMP at 2 time-points, the first prior to surgery (transplantation), and the second 20-28 hours later. At each infusion, the IMP will be followed by a 100ml infusion of 0.9% Sodium Chloride over 15mins.
  Interventions: Drug: Heme Arginate 25 MG/ML
- Placebo Group (Placebo Comparator): Will receive a 100ml infusion of 0.9% Sodium Chloride (placebo) over 30mins. Participants will receive infusions at 2 time-points, the first prior to surgery, and the second 20-28 hours later. At each infusion, the placebo will be followed by a further 100ml infusion of 0.9% Sodium Chloride over 15mins.
  Interventions: Drug: 0.9% Sodium-chloride

INTERVENTIONS:
Drug: Heme Arginate 25 MG/ML — IMP - to be administered at a dose of 3mg/kg to a maximum dose of 250mg over 30 mins. Participants will receive intervention twice during the trial, one on Day 0 (day of transplantation) and then again on D1 (20-28 hours after dose 1).
  Arms: Active Group
Drug: 0.9% Sodium-chloride — Placebo - 100ml of 0.9% Sodium Chloride will be given over 30 mins. Participants will receive intervention twice during the trial, one on Day 0 (day of transplantation) and then again on D1 (20-28 hours after dose 1).
  Arms: Placebo Group

SUMMARY:
Organ shortage for transplant has necessitated use of kidneys from older donors, increasing the chance that the kidney will not work immediately or for as long as expected. The investigators gave the drug heme arginate (HA) to 20 kidney transplant patients in the first 24 hours after transplant, and showed that it may reduce kidney injury and is safe. The investigators plan to conduct a large study recruiting 600 patients to determine whether HA treatment increases the number of kidney transplants that work immediately. If successful, HA may be introduced into clinical practice at the end of this study.

Patients will be invited to take part in the study once listed for a kidney transplant. Further discussions will be had with them when admitted for transplant, and they will be offered the opportunity to participate. Consent will not be taken until the patient is admitted for transplantation. Following consent, participants will be randomised to receive either 2 doses of the study drug, HA, or a salt water solution, one at the time of transplant, and one approximately 24 hours later. Otherwise, treatment will be the same as any other patient undergoing a kidney transplant. Information about recovery from surgery, and specifically about kidney function, will be collected, but will not require additional blood tests. The study period ends after the first 7 days post-transplant, although longer term data will be collected from routine follow up appointments. Participants will be asked to complete a simple quality of life questionnaire 3 times: just before transplant, at approximately one week and three months after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a kidney only transplant, or a dual kidney transplant, from a deceased donor
* At least 18 years of age, no upper limit
* Receiving standard immunosuppression for the individual centre
* (where applicable) Meets co-enrolment criteria outlined in section 4.4 of the protocol

Exclusion Criteria:

* Kidney transplant patients as part of a multi-organ transplant e.g. with pancreas or liver
* Known hypersensitivity to heme arginate
* Unable to give informed consent
* Patients with porphyria, irrespective of whether they have received heme arginate or not, will be excluded
* Previous randomisation into this study (or HOT study)
* Women who are pregnant or lactating
* Kidneys that have undergone Ex-vivo Normothermic Perfusion (EVNP)
* Patients with known liver disease, epilepsy, brain injury or disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Delayed Graft Function | 1 week post transplant
  The incidence of delayed graft function, defined as failure of a spontaneous fall in creatinine of >10% for each 3 consecutive day period in the first week following transplantation, with comparison between the two randomised groups.

SECONDARY OUTCOMES:
Requirement for dialysis | 1 week post transplant
  The number of participants requiring dialysis within the first week post-transplant
Time to functioning graft | 1 week
  The number of days to functioning graft, defined as the spontaneous fall in creatinine of greater than, or equal to 10% over a period of 3 consecutive days in the first 7 days post transplant
Length of hospital stay | 3 months
  The number of days spent in hospital, along with level of care (ward/HDU/ITU), for the index admission (transplantation admission)
Creatinine levels | 3 months
  Serum creatinine levels at 1 and 3 months post-transplant across both randomised groups
Acute rejection | 3 months
  The number of participants with biopsy-proven acute rejection within the first 3 months post-transplant
SF36 Quality of Life | Up to 3 months post transplant
  A comparison of differences between groups in patient reported quality of life using the SF36
Cost per QALY gained | Up to 3 months post transplant
  Using data derived from the SF36 to weight survival for quality of life, Quality Adjusted Life Year (QALY) will be assessed

OTHER OUTCOMES:
1 Year graft survival | 1 year
  Graft survival rates at 1 year post transplant will be obtained from routinely collected data and differences between treatment groups assessed.
1 year recipient survival | 1 year
  Recipient survival rates at 1 year post transplant will be obtained from routinely collected data and differences between treatment groups assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Marson, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - NHS Lothian - Royal Infirmary of Edinburgh, Edinburgh, Lothian
  - Edinburgh Clinical Trials Unit, Usher Institute, University of Edinburgh, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the primary paper, a de-identified individual participant data set will be submitted to a data archive for sharing purposes. Access to this data set will be under a controlled access model in line with ECTU policies at that time.
Supporting Information: Study Protocol, SAP